CLINICAL TRIAL: NCT06856733
Title: Improved Treatment for Patients With Long-term Opioid Therapy for Non-cancer Pain in Primary Care (Opi-Prim)
Brief Title: Improved Treatment for Patients With Long-term Opioid Therapy for Non-cancer Pain in Primary Care
Acronym: Opi-Prim
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala County Council, Sweden (Other Government)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Thomas Kempen, Assistant professor, Uppsala County Council, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Opi-Prim
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Pain; Chronic Pain Management; Primary Care
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control healthcare centres will receive usual care. This may include appointments and treatment by a general practitioner, nurse, physiotherapist and/or psychologist. No pharmacist will be working at the healthcare centre. However, Uppsala County Council does provide centralized medication review services to all primary healthcare centres in Region Uppsala. Any healthcare professional may request a medication review by a pharmacist on a work-from-home basis as part of usual care.
- Intervention (Active Comparator): Phase 1 (investigation and assessment, week 1-3):
  * A medication review focusing on pain, sleep and depression/anxiety disorders by a pharmacist.
  * A thorough pain analysis by a GP according to existing guidelines including duration of pain, pain localization and pain mechanisms.
  * A visit to a physiotherapist for evaluation and assessment of possible treatment regarding physical exercise/physical activities.
  * A visit to a psychologist for diagnostics and treatments regarding psychological and social factors.
  * A visit to a care manager
  Phase 2 (treatment plan, week 3-4):
  - A team consultation with all healthcare personnel involved in Phase 1 including the patient where an individualized rehabilitation plan is made.
  Phase 3 (treatment and follow-up, week 4-24):
  * Implementation of the individualized rehabilitation plan.
  * Frequent follow-up contacts (1 per 1-3 weeks) by phone with an established contact person, i.e. care manager.
  * A second team consultation half-way
  Interventions: Behavioral: Person-centred team-based approach

INTERVENTIONS:
Behavioral: Person-centred team-based approach — Phase 1 (investigation and assessment, week 1-3):
  * A medication review focusing on pain, sleep and depression/anxiety disorders by a pharmacist.
  * A thorough pain analysis by a GP according to existing guidelines including duration of pain, pain localization and pain mechanisms.
  * A visit to a physiotherapist for evaluation and assessment of possible treatment regarding physical exercise/physical activities.
  * A visit to a psychologist for diagnostics and treatments regarding psychological and social factors.
  * A visit to a care manager
  Phase 2 (treatment plan, week 3-4):
  - A team consultation with all healthcare personnel involved in Phase 1 including the patient where an individualized rehabilitation plan is made.
  Phase 3 (treatment and follow-up, week 4-24):
  * Implementation of the individualized rehabilitation plan.
  * Frequent follow-up contacts (1 per 1-3 weeks) by phone with an established contact person, i.e. care manager.
  * A second team consultation half-way
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to reduce inappropriate long term opioid treatment (LTOT) and to optimize pain management in patients with LTOT for chronic non-cancer pain in primary care through a new person-centred and team-based approach. The main question it aims to answer is:

What are the effects of a new person-centred and team-based approach on pain interference in patients with LTOT for chronic non-cancer pain in primary care?

Researchers will compare a new person-centred and team-based approach to usual care to see if pain interference is lower.

Participants will receive a person-centred team-based treatment consisting of:

* Phase 1 (investigation and assessment, week 1-3): A medication review, pain analysis and other assessments through separate visits to a pharmacist, general practitioner, physiotherapist, psychologist and care manager
* Phase 2 (treatment plan, week 3-4): A team consultations with all healthcare personnel involved in Phase 1 including the patient where an individualized rehabilitation plan is made based.
* Phase 3 (treatment and follow-up, week 4-24): Implementation of the individualized rehabilitation plan with frequent follow-up contacts (1 per 1-3 weeks) by phone with the care manager.

DETAILED DESCRIPTION:
The evidence for prescribing opioids to patients suffering from chronic non-cancer pain is weak, and using opioids in these circumstances is questionable. Swedish primary health care is responsible for about one-third of all first-time opioid prescriptions and has the highest rate of prescription renewals for opioids. The decision for long-term opioid therapy (LTOT) should rest on an accurate pain analysis and should result in an individualized assessment where the risks of LTOT are set against the impact on quality of life that living with long-term pain entails. Multi-professional interventions and a person-centered approach are recommended for chronic non-cancer pain. Although pharmacists in primary health care have been established internationally with successful examples related to LTOT, their role in Swedish primary care and the management of chronic non-cancer pain remains to be studied. Currently, it is unclear which interventions are effective in reducing inappropriate LTOT and which alternative interventions are suitable for patients who are currently receiving LTOT. The involvement of a care manager in the patient´s care has shown promising results regarding quality of care for other long-term conditions, for example depresssion. In Region Uppsala, clinical pharmacists havte recently been employed in primary health care, but it is unclear what their tasks and responsibilities are and how to best make use of their competence. It is therefore relevant and justified to investigate a new person-centered team-based approach including care manager and pharmacist to optimize the management of pain in patients with chronic non-cancer pain in Swedish primary care. This project aims to reduce inappropriate LTOT and optimize pain management in patients with LTOT for chronic non-cancer pain in primary care through a new person-centered and team-based approach.

Primary objective:

To investigate the effects of a new person-centred and team-based approach on pain interference in patients with LTOT for chronic non-cancer pain in primary care

Trial design and setting:

This study is a controlled before-and-after study that has been designed, and will be reported, according to the CONSORT guidelines. Participation will be during 52 weeks (12 months).

This study will be conducted at eight healthcare centres in Region Uppsala. At four of the healthcare centres, a new person-centred team-based treatment model including pharmacists (intervention) will be implemented. Prerequisites for these healthcare centres are the accessibility of at least one person of each healthcare profession: pharmacist, general practitioner (GP), psychologist (or social worker) and physiotherapist, where one of these (or a rehabilitation coordinator or a nurse) takes the role of care manager. Healthcare personnel will receive special training in managing patients with chronic pain before the study. In addition, four control healthcare centres without a pharmacist will be matched with the intervention healthcare centres according to geographic area (urban, suburban, rural), socioeconomical setting and the size of the centres (number of listed patients). No specific efforts of implementation will be made in these control centres.

Prior to the full trial, a feasibility study will be conducted at one intervention centre and one control centre with 12 weeks follow-up per participant.

ELIGIBILITY:
Inclusion Criteria:

* Having received the equivalent of 90 days or more prescription of opioids for chronic pain made by the general practitioner during the recent 12 months
* Able to speak Swedish or English

Exclusion Criteria:

* Having been referred to a pain clinic (either at hospital or multimodal rehabilitation in primary care) within the last 6 months
* No current opioid use, severe cognitive dysfunction, e.g., suicidal ideation, psychotic symptoms, or dementia, that prevents informed consent.
* Using their opioids for cancer pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain interference | The primary outcome measure will be the difference in mean pain interference after 6 months.
  Measured with the Brief Pain Inventory - Short Form (BPI-SF), question number 9 a-g. Scale: 0-10. Higher score is worse.

SECONDARY OUTCOMES:
Pain intensity | After 3, 6 and 12 months
  Measured with the Brief Pain Inventory - Short Form (BPI-SF), question number 3-8. Scale: 0-10. Higher score is worse
Symptoms of depression | After 3, 6 and 12 months
  Measured with the Patient Health Questionnaire-9 (PHQ-9). Scale: 0-27. Higher score is worse
Symptoms of anxiety | After 3, 6 and 12 months
  Measured with the General Anxiety disorder-7 (GAD-7). Scale: 0-27. Higher score is worse
Patient satisfaction | After 3, 6 and 12 months
  Measured with the Patients´ Global impression of Change (PGIC). Scale: 0-6. Higher score is worse
Quality of life according to the 5-level EuroQol 5D | After 3, 6 and 12 months
  Measured with the 5-level EuroQol 5D (EQ-5D-5L). Scale: 1-5 per dimension. Higher score is worse.
Opioid use | After 3, 6 and 12 months
  Measured with as morphine equivalents: in mg.
Symptoms of withdrawal | After 3, 6 and 12 months
  Measured with the Short Opioid Withdrawal Scale (SOWS). Scale: 0-40. Higher score is worse
Pain interference | After 3 and 12 months
  Measured with the Brief Pain Inventory - Short Form (BPI-SF), question number 9 a-g. Scale: 0-10. Higher score is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Region Uppsala, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT06856733/Prot_000.pdf